CLINICAL TRIAL: NCT00308841
Title: Anesthetic Efficacy of Intrauterine Lidocaine for Removal of a "Lost" Intrauterine Device
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Suleyman Demirel University (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: B.30.2.SDÜ.0.01.00.01.301.01
Record Dates: First submitted 2006-03-29; First posted 2006-03-30 (Estimated); Last update posted 2008-10-20 (Estimated); Status verified 2005-09

CONDITIONS: "Lost" IUD
Keywords: Objective: To evaluate the efficacy of intrauterine lidocaine instillation in reducing patient discomfort during the removal of a "lost" IUD
MeSH Terms: interventions — Lidocaine; Pharmaceutical Preparations

INTERVENTIONS:
Drug: Lidocaine (drug)

SUMMARY:
Objective: To evaluate the efficacy of intrauterine lidocaine instillation in reducing patient discomfort during the removal of a "lost" intrauterine device (IUD).

Methods: This double-blinded, randomized, placebo-controlled trial included 68 women who underwent removal procedure for a "lost" IUD. Thirty-four women were allocated to the lidocaine group and 34 to the saline group. The main outcome measure was the intensity of pain during, immediately after, and 20 minutes after the procedure, assessed by a visual analog scale. Statistical analysis was performed using Friedman's test with Bonferroni correction, Student's t test, and 2.

ELIGIBILITY:
Inclusion Criteria:

patients undergoing a minor gynecologic procedure for removal of a "lost" IUD.

Exclusion Criteria:

women with a history of cervical stenosis, known allergy to lidocaine, pregnancy, acute cervicitis

Sex: Female
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Güney, M.D, Principal Investigator — SDU
Locations (1):
- Süleyman Demirel University, School of Medicine, Isparta, Turkey (Türkiye)

REFERENCES:
- [Result] Guney M, Oral B, Mungan T. Efficacy of intrauterine lidocaine for removal of a "lost" intrauterine device: a randomized, controlled trial. Obstet Gynecol. 2006 Jul;108(1):119-23. doi: 10.1097/01.AOG.0000223201.42144.80. PMID 16816065